CLINICAL TRIAL: NCT07326176
Title: Evaluating Pathophysiological Mechanisms of Acute and Chronic Heat Stress on Maternal and Fetal Health
Acronym: GaHPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Leonidas G. Ioannou, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GaHPS; 227176/Z/23/Z (Other Grant/Funding Number: Wellcome)
Record Dates: First submitted 2025-12-10; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Thermally Neutral Condition With Light-intensity Work; Thermally Neutral Condition With Moderate-intensity Work; Warm Condition With Light-intensity Work; Warm Condition With Moderate-intensity Work
Keywords: heat stress; heat strain
MeSH Terms: conditions — Heat Stress Disorders | interventions — Hot Temperature

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Temperate-Light (Other): Participants were exposed to a temperate environment (20 °C, 45% relative humidity, shaded) for a 3-hour protocol consisting of 1 hour passive seated exposure, 1 hour of light-intensity treadmill walking (alternating between 2 and 3 METs [Metabolic Equivalents] every 10 minutes), and 1 hour seated recovery.
  Interventions: Other: Heat and Physical Work Exposure Protocol
- Temperate-Moderate (Other): Participants were exposed to a temperate environment (20 °C, 45% relative humidity, shaded) for a 3-hour protocol consisting of 1 hour passive seated exposure, 1 hour of moderate-intensity treadmill walking (alternating between 3 and 4 METs every 10 minutes), and 1 hour seated recovery.
  Interventions: Other: Heat and Physical Work Exposure Protocol
- Warm-Light (Other): Participants were exposed to a warm environment (30 °C, 45% relative humidity, shaded) for a 3-hour protocol consisting of 1 hour passive seated exposure, 1 hour of light-intensity treadmill walking (alternating between 2 and 3 METs every 10 minutes), and 1 hour seated recovery.
  Interventions: Other: Heat and Physical Work Exposure Protocol
- Warm-Moderate (Other): Participants were exposed to a warm environment (30 °C, 45% relative humidity, shaded) for a 3-hour protocol consisting of 1 hour passive seated exposure, 1 hour of moderate-intensity treadmill walking (alternating between 3 and 4 METs every 10 minutes), and 1 hour seated recovery.
  Interventions: Other: Heat and Physical Work Exposure Protocol

INTERVENTIONS:
Other: Heat and Physical Work Exposure Protocol — A controlled 3-hour environmental chamber protocol consisting of 1 hour of passive seated exposure, 1 hour of treadmill walking at prescribed light or moderate intensities (alternating between 2-3 METs or 3-4 METs every 10 minutes), and 1 hour of seated recovery. Each session was conducted under either temperate (20 °C, 45% relative humidity, shaded) or warm (30 °C, 45% relative humidity, shaded) environmental conditions. Environmental settings, workload intensity, and timing were standardized across all participants.

SUMMARY:
This study examined the effects of environmental heat and physical work on maternal thermoregulation and fetal physiology in late pregnancy. Twenty-four healthy pregnant women at 28-32 weeks of gestation completed four randomized and counterbalanced 3-hour experimental scenarios combining two thermal conditions (temperate 20 °C and warm 30 °C, both at 45% relative humidity, shaded) and two physical workload intensities (light and moderate treadmill walking). Each scenario included 1 hour of passive seated exposure, 1 hour of treadmill walking, and 1 hour of seated recovery. Maternal thermoregulatory, cardiovascular, perceptual, and hydration responses were monitored continuously, while fetal heart rate and Doppler-derived indices of uterine, umbilical, and middle cerebral artery blood flow were assessed at baseline, end of passive exposure, end of work, and end of recovery. The aims of the study were: (1) to characterize maternal physiological and perceptual responses to heat exposure and physical work; (2) to determine whether maternal physiological heat strain directly affects fetal cardiovascular strain and maternal-fetal hemodynamics; and (3) to examine whether maternal characteristics, particularly body mass index and age, influence maternal thermoregulatory responses and fetal susceptibility to heat stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women between 28 and 32 weeks of gestation
* Singleton pregnancy
* Habitually heat-acclimatized, defined as daily exposure to outdoor environmental conditions equal to or warmer than those used in the study
* Able to perform treadmill walking at light and moderate intensities
* Willing and able to attend all laboratory sessions
* Provided written informed consent
* Age 18 years or older

Exclusion Criteria:

* Multiple pregnancy (e.g., twins, triplets)
* Chronic medical conditions, including but not limited to:

  * Hypertension
  * Diabetes
  * HIV
* Obstetric complications, including:

  * Pre-eclampsia
  * Severe anemia
* Acute infections, including urinary tract infection
* Any contraindication to exercise based on the Physical Activity Readiness for Pregnancy (PARmed-X for Pregnancy) checklist
* Inability to comply with the study procedures or scheduled visits
* Any condition deemed by investigators to compromise participant safety or data integrity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 24 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Maternal Core Body Temperature | Continuously recorded throughout each 3-hour experimental session (baseline, 1-hour passive exposure, 1-hour physical work, and 1-hour recovery).
  Core body temperature continuously assessed using an ingestible telemetric temperature capsule to quantify maternal thermoregulatory responses to different combinations of environmental heat (20 °C vs 30 °C) and physical workload (light vs moderate).
Maternal Physiological Strain Index | Continuously calculated throughout each 3-hour experimental session (baseline, passive exposure, physical work, and recovery).
  Physiological Strain Index (0-10 scale) calculated from core body temperature and heart rate to quantify overall maternal physiological heat strain under different environmental and workload combinations.
Fetal Heart Rate | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Fetal heart rate assessed using obstetric ultrasound to evaluate fetal cardiovascular responses to maternal exposure to different environmental temperatures and physical workload intensities.
Uterine Artery Pulsatility Index (PI) | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Pulsatility Index of the left and right uterine arteries measured by Doppler ultrasound to assess uteroplacental vascular resistance under different environmental and workload conditions.
Uterine Artery Resistive Index (RI) | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Resistive Index of the left and right uterine arteries measured by Doppler ultrasound to assess uteroplacental vascular resistance under different environmental and workload conditions.
Umbilical Artery Pulsatility Index | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Pulsatility Index of the umbilical artery measured by Doppler ultrasound to evaluate fetoplacental blood flow in response to maternal heat exposure and physical work.
Umbilical Artery Resistive Index | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Resistive Index of the umbilical artery measured by Doppler ultrasound to evaluate fetoplacental blood flow in response to maternal heat exposure and physical work.
Middle Cerebral Artery Pulsatility Index | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Pulsatility Index of the fetal middle cerebral artery measured by Doppler ultrasound to assess fetal cerebral vascular responses to maternal heat strain.
Middle Cerebral Artery Resistive Index | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Resistive Index of the fetal middle cerebral artery measured by Doppler ultrasound to assess fetal cerebral vascular responses to maternal heat strain.
Composite Maternal-Fetal Hemodynamic Ratios (cerebroplacental ratio) | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Cerebroplacental ratio calculated using artery Doppler measurements to characterize maternal-fetal hemodynamics and fetal strain under different environmental and workload conditions.
Composite Maternal-Fetal Hemodynamic Ratios (cerebrouterine PI ratio) | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Cerebrouterine PI ratio calculated using artery Doppler measurements to characterize maternal-fetal hemodynamics and fetal strain under different environmental and workload conditions.
Composite Maternal-Fetal Hemodynamic Ratios (Uteroplacental:cerebral PI ratio) | Each 3-hour session: 0 min (baseline), 60 min (end of passive exposure), 120 min (end of physical work), 180 min (end of recovery).
  Uteroplacental:cerebral PI ratio calculated using artery Doppler measurements to characterize maternal-fetal hemodynamics and fetal strain under different environmental and workload conditions.

SECONDARY OUTCOMES:
Maternal Skin Temperature | Continuously recorded throughout each 3-hour experimental session (baseline, passive exposure, physical work, and recovery).
  Skin temperature measured at four body sites (chest, upper arm, thigh, lower leg) using iButton sensors and expressed as a weighted mean skin temperature to characterize peripheral thermal responses to environmental heat and physical work.
Maternal Heart Rate | Continuously recorded throughout each 3-hour experimental session (baseline, passive exposure, physical work, and recovery).
  Maternal heart rate measured using a chest-strap heart rate monitor to assess cardiovascular strain across different environmental (20 °C vs 30 °C) and workload (light vs moderate) conditions.
Maternal Local Sweat Rate | Continuously recorded throughout each 3-hour experimental session (baseline, passive exposure, physical work, and recovery).
  Local sweat rate measured over the trapezius muscle using a ventilated capsule technique, adjusted for skin area, to quantify sweating responses to environmental heat and physical work.
Maternal Skin Blood Flow | Continuously recorded throughout each 3-hour experimental session (baseline, passive exposure, physical work, and recovery).
  Skin blood flow assessed using laser Doppler flowmetry at the finger and forearm to characterize peripheral vasodilation in response to environmental heat exposure and physical work.
Maternal Arterial Blood Pressure | Measured at baseline and every 30 minutes during each 3-hour experimental session.
  Systolic, diastolic, and mean arterial blood pressure measured intermittently using a standard automated sphygmomanometer to evaluate cardiovascular responses to environmental heat and physical work.
Thermal Sensation | Measured at baseline and every 30 minutes throughout each 3-hour experimental session (passive exposure, physical work, and recovery).
  Thermal sensation assessed using a 9-point scale ranging from -4 (extremely cold) to +4 (extremely hot) to quantify participants' perceived body temperature during exposure to different environmental heat and physical workload conditions.
Thermal Comfort | Measured at baseline and every 30 minutes throughout each 3-hour experimental session (passive exposure, physical work, and recovery).
  Thermal comfort assessed using a 10-point scale ranging from 1 (comfortable) to 10 (extremely uncomfortable) to evaluate subjective comfort during environmental heat exposure and physical work.
Rating of Perceived Exertion (RPE) | Measured at baseline and every 30 minutes throughout each 3-hour experimental session (passive exposure, physical work, and recovery).
  Perceived exertion assessed using the Borg 6-20 scale to quantify subjective physical effort during treadmill walking under different environmental and workload conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Ioannou, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Dept. of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of the data collected from pregnant women and their fetuses and the potential risk of re-identification. De-identified, non-trackable aggregated data supporting the main study findings will be made available after publication.

REFERENCES:
- [Background] Bonell A, Sonko B, Badjie J, Samateh T, Saidy T, Sosseh F, Sallah Y, Bajo K, Murray KA, Hirst J, Vicedo-Cabrera A, Prentice AM, Maxwell NS, Haines A. Environmental heat stress on maternal physiology and fetal blood flow in pregnant subsistence farmers in The Gambia, west Africa: an observational cohort study. Lancet Planet Health. 2022 Dec;6(12):e968-e976. doi: 10.1016/S2542-5196(22)00242-X. PMID 36495891
- [Background] Bonell A, G Ioannou L, Sesay A, A Murray K, Bah B, Jeffries D, E Moore S, Vicero-Cabrera A, S Maxwell N, E Hirst J, Tan C, Saucy A, Watters D, Sonko B, Okoh E, Idris Y, Oluwatosin Adefila W, Manneh J, Leigh-Nabou M, Bojang S, Flouris A, Haines A, Prentice A, N Sferruzzi-Perri A. Study protocol for an observational cohort study of heat stress impacts in pregnancy in The Gambia, West Africa. Wellcome Open Res. 2025 Feb 7;9:624. doi: 10.12688/wellcomeopenres.23172.2. eCollection 2024. PMID 39925648
- See also: Related Info — https://www.lshtm.ac.uk/research/centres-projects-groups/gambia-heat-in-pregnancy-study